CLINICAL TRIAL: NCT01683695
Title: A Randomized, Double-blind, Parallel, Placebo-controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Effect of AMG 557 in Systemic Lupus Erythematosus (SLE) Subjects With Active Lupus Arthritis
Brief Title: Safety Study of AMG 557 in Subjects With Lupus Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101103
Record Dates: First submitted 2012-03-14; First posted 2012-09-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Lupus Arthritis, Systemic Lupus Erythematosus
Keywords: Lupus Arthritis, Systemic Lupus Erythematosus, AMG 557, Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — AMG 557

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 557 (Active Comparator): All will receive AMG 557 on Day 1, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113, Day 127, Day 141 and Day 155.
  Interventions: Drug: AMG 557
- AMG 557 Matching Placebo (Placebo Comparator): All will receive AMG 557 on Day 1, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113, Day 127, Day 141 and Day 155.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: AMG 557 — AMG 557 will be administered as subcutaneous injections in the anterior abdomen of the subjects.
  Arms: AMG 557
Drug: Matching Placebo — Placebo will be administered as subcutaneous injections in the anterior abdomen of the subjects.
  Arms: AMG 557 Matching Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel, placebo-controlled, multiple dose study that will enroll approximately 40 systemic lupus erythematosus subjects with active lupus arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE for at least 6 months as defined by the most recent American College of Rheumatology criteria
* Presence of lupus related inflammatory arthritis with at least four tender and four swollen joints; and Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) ≥ 6 at screening;
* Other inclusion criteria may apply.

Exclusion Criteria:

* Presence or history of vasculitis, and presence or history of active lupus nephritis requiring therapy within the last 3 years
* Any disorder (including psychiatric), condition, clinically significant disease, disease activity related to SLE
* Positive for HIV antibodies, hepatitis B surface antigen or anti-HBc, or hepatitis C antibodies
* Known residential exposure to an individual with tuberculosis or positive Quantiferon test or PPD test at screening
* Men and women of reproductive potential, unwilling to practice a highly effective method of birth control for the duration of the study
* Other exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events, vital signs, physical examinations, clinical laboratory tests, ECGs, and the incidence of binding and neutralizing antibodies to AMG 557. | 330 days, including a 21-day screening period
Lupus Arthritis Response Rate | Day 169
  Defined by: 1) achieving at least a 50% decrease in the combined tender and swollen joint count compared to baseline at Day 169; 2) achieving one letter improvement in the Musculoskeletal System BILAG at Day 169 compared to baseline; 3) reduction in and maintenance of prednisone (or its equivalent) dose to ≤ 50% of baseline corticosteroid dose (Day 1 predose) or ≤ 7.5 mg/day, whichever is lower, from Day 85 to Day 169 in subjects not treated with immunosuppressants at baseline, or reduction in and maintenance of prednisone (or its equivalent) dose to ≤ 7.5 mg/day from Day 85 to Day 169 and discontinuation of immunosuppressants by Day 29 in subjects treated with immunosuppressants at baseline

SECONDARY OUTCOMES:
Proportion of subjects achieving a) one letter improvement; and b) 'C' or better score in the Musculoskeletal system from BILAG index at Day 169 compared to baseline, by treatment group. | Day 169
Percentage change in the tender and swollen joint counts at Day 169 relative to baseline. | Day 169
Proportion of subjects achieving reduction in and maintenance ≤ 7.5 mg/day of prednisone (or equivalent) from Day 85- Day 169 and discontinuation of immunosuppressants by Day 29 in subjects treated with immunosuppressants at baseline. | Days 85-169
Proportion of subjects achieving reduction in and maintenance of prednisone (or its | Days 85-169
Physician Global Assessment of Disease Activity (PGADA). | 330 days, including a 21-day screening period
Subject Global Assessment of Disease Activity (SGADA). | 330 days, including a 21-day screening period
Serum PK profile of AMG 557 after multiple dose administrations. | 330 days, including a 21-day screening period
Proportion of subjects who discontinued immunosuppressants by Day 29 in subjects | Day 29
Cumulative dose of prednisone (or its equivalent) from Day 85 to Day 169. | Day 85 to Day 169

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, San Leandro, California
  - Research Site, Danbury, Connecticut
  - Research Site, Manhasset, New York
- Research Site, St Leonards, New South Wales, Australia
- Research Site, Odense, Denmark
- Research Site, Lille, France
- Research Site, Berlin, Germany
- Malaysia (2):
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kuching, Sarawak
- Research Site, Taipei, Taiwan
- United Kingdom (2):
  - Research Site, Birmingham
  - Research Site, London

REFERENCES:
- [Derived] Cheng LE, Amoura Z, Cheah B, Hiepe F, Sullivan BA, Zhou L, Arnold GE, Tsuji WH, Merrill JT, Chung JB. Brief Report: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multiple-Dose Study to Evaluate AMG 557 in Patients With Systemic Lupus Erythematosus and Active Lupus Arthritis. Arthritis Rheumatol. 2018 Jul;70(7):1071-1076. doi: 10.1002/art.40479. Epub 2018 May 25. PMID 29513931
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com